CLINICAL TRIAL: NCT05621096
Title: Feasibility of Low Dose Radiation as Bridging Therapy for Lisocabtagene Maraleucel in Relapsed B-Cell Non-Hodgkin Lymphoma
Brief Title: Low Dose Radiation as Bridging Therapy in Relapsed B-Cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0770-22-FB
Record Dates: First submitted 2022-10-27; First posted 2022-11-17 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; Follicular Lymphoma; Mediastinal Large B-cell Lymphoma; Indolent B-Cell Non-Hodgkin Lymphoma; Relapsed Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — Receptors, Chimeric Antigen; Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm (Experimental): Subjects will receive 4 gray (Gy) radiation in 2 fractions in the bridging period following lymphocyte pheresis, prior to lymphodepleting chemotherapy and chimeric antigen receptor (CAR) T-cell infusion. Post CAR T-cell infusion radiation therapy will be allowed as determined by study investigator but prespecified at time of radiation oncology consultation.
  Interventions: Radiation: Bridging radiation therapy; Biological: Liso-cel; Radiation: Post-infusion radiation

INTERVENTIONS:
Radiation: Bridging radiation therapy — Days -20 to -7: Patients will receive 2 fractions of 2 gray (Gy) for a total of 4 Gy received.
Biological: Liso-cel — Day 0: Patients will receive an infusion of liso-cel CAR T-cell product.
  Prior to the liso-cell infusion (Days -5 to -3), patients will receive lymphodepleting chemotherapy using fludarabine 30mg/m2 and cyclophosphamide 300mg/m2 per institutional standard procedures.
  Other Names: Chimeric antigen receptor (CAR) T-cell product
Radiation: Post-infusion radiation — Days 30 to 80: Patients eligible for post-infusion radiation will receive a total dose of up to 32 Gy.

SUMMARY:
The goal of this clinical trial is to learn about treatment for people with B-cell lymphoma that did not respond to treatment or that has gotten worse after treatment. The aim of this trial is to answer the following questions:

* If it is realistic to give people radiation treatment before they receive a chimeric antigen receptor (CAR) T-cell treatment for their cancer
* If it is safe to give people radiation treatment before they receive a CAR T-cell treatment for their cancer

DETAILED DESCRIPTION:
This is a pilot study to evaluate the feasibility of low-dose radiation therapy in the bridging period between chimeric antigen receptor (CAR) T-cell collection, manufacturing, and infusion (vein-to-vein) in patients with relapsed and refractory aggressive B-cell lymphoma.

Emerging cellular immunotherapies including CAR T-cell therapy have produced remarkable outcomes for this population. The Food and Drug Administration (FDA) has recently approved lisocabtagene maraleucel (liso-cel) for the management of people with relapsed and refractory B-cell lymphoma. Unfortunately, many patients undergoing liso-cel infusion will suffer progression or relapse with devastating consequences. The object of this study is to identify a novel means to enhance liso-cel activity to improve overall outcomes. The investigators hypothesize that the addition of radiation therapy targeting selected sites as bridging therapy prior to lymphodepleting chemotherapy and liso-cel infusion will be effective at improving responses for patients with relapsed and refractory B-cell lymphoma.

Results from this study will provide key justification to expand this therapeutic approach into a larger phase II clinical trial powered to examine the efficacy of this approach.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven relapsed or progressive diffuse large B-cell lymphoma (DLBCL), high-grade B-cell lymphoma, primary mediastinal B-cell lymphoma, grade 3B follicular lymphoma, or DLBCL arising from indolent lymphoma meeting an FDA-approved (Food and Drug Administration-approved) indication for liso-cel infusion
2. Presence of disease on imaging including at least one disease site safe for radiation as determined by treating radiation oncologist
3. Willingness to participate in clinical trial and provide informed consent
4. Adequate organ function as assessed by standard institution protocols and United States (US) prescribing information label for comorbidities, heart, and lung function to undergo FDA-approved CAR T-cell therapy as determined by institution
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
6. Age 19 years or older, there is no upper limit to the age

Exclusion Criteria:

1. Subject is unsafe for radiation therapy as determined by investigator and/or radiation oncologist
2. Diagnosis is primary central nervous system (CNS) lymphoma (secondary CNS lymphoma with additional systemic site is allowed)
3. Requirement for concurrent high dose methotrexate
4. Secondary active malignancy that has not been in remission for at least 2 years. This excludes non-melanoma skin cancer, definitively treated stage 1 solid tumor with low risk or recurrence, and curatively treated localized prostate cancer.
5. Pregnant or nursing women
6. Uncontrolled medical, psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol, as determined by investigator
7. Unwillingness to follow procedures required in the protocol
8. Inadequate organ or hematologic conditions that prohibit the use of lymphodepleting chemotherapy
9. Use of lymphoma-directed therapy within 14 days of T-cell pheresis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention in the proposed study population | Up to 90 days
  The percentage of subjects who receive a chimeric antigen receptor (CAR) T-cell infusion after receiving bridging radiation therapy. A one-sided Binomial test will be conducted to assess whether acceptable percentage (>70% vs <70%) of patients receive CAR T-cell perfusion after undergoing the radiation therapy.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events to assess the safety of the proposed intervention | Up to 120 days
  Assessed via the incidence of combined Grade 3 and 4 cytokine release syndrome (CRS) or immune effector cell associated neurotoxicity syndrome (ICANS) events as measured by the American Society of Transplant and Cellular Therapy (ASTCT) consensus grading. The grading scale ranges from Grade 1 to 4, with a higher grade indicating a worse outcome. Assessed from the cumulative CRS and ICANS events occurring by the D+30 visit.
Evaluate the response to the study intervention of radiation and CAR T-cell therapy | Up to 190 days
  Response rate will be assessed via PET/CT (positron emission tomography/computed tomography) using Lugano criteria. Overall response rate (ORR) will be defined as the proportion of patients with either a complete response (CR) or a partial response (PR) at D+100. For ORR, CR, and PR: two-sided exact binomial 95% confidence interval of response rate will be constructed to assess the precision of the point estimate.
Evaluate progression-free survival (PFS) following the study intervention | Measured from first day of apheresis to death or disease progression, whichever comes first, up to two years
  PFS will be measured using the Kaplan-Meier method. Disease progression will be measured according to clinical and imaging assessment (Lugano criteria) and will require biopsy confirmation.
Evaluate duration of response (DOR) following CAR T-cell therapy | Up to 2 years
  DOR will be summarized using the Kaplan-Meier method, but only for patients who have achieved a response of at least partial response. DOR is defined by time of first response (D+30 visit) to disease progression, start of new antineoplastic therapy due to efficacy concerns, or death from any cause.
Evaluate overall survival (OS) following study intervention | Up to 2 years
  OS will be analyzed by the Kaplan-Meier method. Subjects alive at last follow up will be censored.
Evaluate the rate of prolonged cytopenias following the intervention | Up to 190 days
  The rate of prolonged cytopenias will be measured as a proportion of subjects with Grade 3 or higher hematologic toxicities per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria at the D+100 visit. The 95% confidence interval will be estimated.
  The CTCAE v5.0 grading system ranges from Grade 0 to 5, with a higher grade indicating a worse outcome.
Monitor overall safety and toxicity of the intervention | Up to 270 days
  Toxicity will be graded using CTCAE v5.0 guidelines. Grade 3 or higher toxicities will be tabulated using percentages at each follow up. The Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grading system ranges from Grade 0 to 5, with a higher grade indicating a worse outcome.
Monitor Cytokine release syndrome (CRS) and Immune effector cell-associated neurotoxicity syndrome (ICANS) toxicity events | Up to 270 days
  Cytokine release syndrome (CRS) and Immune effector cell-associated neurotoxicity syndrome (ICANS) toxicity events will be collected for all grades as measured by American Society for Transplantation and Cellular Therapy (ASTCT) consensus criteria.
  The ASTCT consensus criteria grading system ranges from Grade 1 to 4, with a higher grade indicating a worse outcome.

OTHER OUTCOMES:
Prospectively bank serum and peripheral blood mononuclear cells (PBMCs) | Up to 270 days
  Storage for subsequent correlative analyses in future research. No analysis plan is provided.
Prospectively bank stool samples for future gut microbiome exploratory analyses | Up to 270 days
  Sample storage at indicated timepoints. No specific analysis is intended on this protocol
Evaluate in-field versus out-of-field disease progression following radiation therapy | Up to 270 days
  Proportion of individual disease sites with local progression by Lugano criteria defined by within the treated radiation field versus outside the treated radiation field

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R D'Angelo, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No